CLINICAL TRIAL: NCT05316155
Title: Phase 1/2 Study of Erdafitinib Intravesical Delivery System (TAR-210) in Participants With Non-Muscle-Invasive or Muscle-Invasive Bladder Cancer
Brief Title: Study of Erdafitinib Intravesical Delivery System for Localized Bladder Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109115; 42756493BLC1003 (Other: Janssen Research & Development, LLC); 2021-004144-22 (EudraCT Number); 2023-506265-65-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Non-Muscle Invasive Bladder Neoplasms
Keywords: Non-Muscle Invasive Bladder Cancer (NMIBC); Muscle Invasive Bladder Cancer (MIBC)
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — erdafitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Dose Escalation (Experimental): Participants with recurrent, bacillus Calmette-Guerin (BCG)-experienced high risk papillary-only Non-Muscle-Invasive Bladder Cancer (NMIBC), refusing or ineligible for radical cystectomy or with recurrent, intermediate-risk NMIBC will receive Erdafitinib Intravesical Delivery System. The dose will be escalated to determine preliminary recommended phase 2 dose(s) (RP2D[s]) for Part 2.
  Interventions: Drug: Erdafitinib Intravesical Delivery System
- Part 2: Dose Expansion (Experimental): Participants in each of 5 disease-specific NMIBC or MIBC cohorts may be enrolled at one or more dose levels that have been determined to be safe in Part 1.
  Interventions: Drug: Erdafitinib Intravesical Delivery System
- Part 3: RP2D Dose Expansion (Experimental): Participants in 2 of the disease-specific NMIBC cohorts (cohorts 1 and 3) may be enrolled at RP2D to determine the safety, evaluate PK and preliminary clinical activity.
  Interventions: Drug: Erdafitinib Intravesical Delivery System
- Part 4: Phase 2 Expansion (Experimental): Participants with recurrent IR-NMIBC will be enrolled in this part to further evaluate the safety, efficacy, and PK of the selected RP2D.
  Interventions: Drug: Erdafitinib Intravesical Delivery System

INTERVENTIONS:
Drug: Erdafitinib Intravesical Delivery System — Erdafitinib intravesical delivery system will be administered.
  Other Names: JNJ-42756493

SUMMARY:
The purpose of the study in Part 1 (dose escalation) and in Part 2 (dose expansion) is to determine the recommended Phase 2 dose(s) (RP2D[s]) and evaluate preliminary clinical efficacy. Part 3 (dose expansion) will confirm safety and preliminary clinical activity at the RP2D. Part 4 (RP2D expansion; MoonRISe-2) will assess the overall complete response (CR) in participants with intermediate-risk-non-muscle invasive bladder cancer (IR-NMIBC; means the cancer cells are only in the bladder's inner lining).

DETAILED DESCRIPTION:
Bladder cancer is one of the most common malignancy worldwide, and non-muscle invasive (NMIBC) requires intensive regimens of frequent monitoring and local resection (transurethral resection of bladder [TURBT]). This study enrolls participants with non-muscle invasive or muscle invasive bladder cancer with activating fibroblast growth factor receptor (FGFR) mutations or fusions. Erdafitinib is a pan-FGFR inhibitor with demonstrated clinical activity when administered orally in patients with solid tumors, including bladder cancer, with FGFR genetic alterations. The Erdafitinib intravesical delivery system is designed to provide release of Erdafitinib in the bladder to treat localized bladder cancer, while reducing systemic toxicities. The study consists of a screening phase, a treatment phase, and a follow-up phase. Total duration of the study is approximately up to 7 years 4 months.

ELIGIBILITY:
Inclusion Criteria:

Parts 1-3:

* Muscle-invasive or recurrent, non-muscle-invasive urothelial carcinoma of the bladder
* For selected Cohorts: Activating tumor pan-fibroblast growth factor receptor (FGFR) mutation or fusion, as determined by local or central testing, approved by the sponsor prior to the start of study treatment. Local tissue-based results (if already existing) from next-generation sequencing (NGS) or polymerase chain reaction (PCR) tests performed in Clinical Laboratory Improvement Amendments (CLIA) -certified or equivalent laboratories, or results from commercially available PCR or NGS tests
* Cohorts 1 and 2: Bacillus Calmette-Guérin (BCG) experienced, or participants with no BCG experience because BCG was not available as a treatment option in the participant's location within the previous 2 years and is currently unavailable. Participants who received an abbreviated course of BCG due to toxicity are still eligible
* Cohort 1 only: Refuses or is not eligible for radical cystectomy (RC)
* Cohorts 2 and 4: Willing and eligible for RC

Part 4:

* Have histologically confirmed diagnosis of recurrent Intermediate-risk-non-muscle invasive bladder cancer (IR-NMIBC) Ta LG tumors
* Must not have undergone tumor debulking or selective ablation of visible lesions; partial tumor biopsy to confirm diagnosis and provide tissue for biomarker testing is permitted as long as remaining tumor is at least 5 millimeter (mm) in size
* Must submit tissue and urine for FGFR testing
* Can have a prior or concurrent second malignancy which natural history or treatment is unlikely to interfere with any study endpoints of safety or the efficacy of the study treatment

Exclusion Criteria:

Parts 1-3:

* Concurrent extra-vesical (that is, urethra, ureter, renal pelvis) transitional cell carcinoma of the urothelium
* Prior treatment with an pan-fibroblast growth factor receptor (FGFR) inhibitor
* Received pelvic radiotherapy <=6 months prior to the planned start of study treatment. If received pelvic radiotherapy greater than (>)6 months prior to the start of study treatment, there must be no cystoscopic evidence of radiation cystitis
* Presence of any bladder or urethral anatomic feature that in the opinion of the investigator may prevent the safe use of Erdafitinib intravesical delivery system
* Indwelling urinary catheter. Intermittent catheterization is acceptable

Part 4:

* Histologically confirmed diagnosis of T1 NMIBC, HR NMIBC (HG/G2 or HG/G3 or CIS) or MIBC, locally advanced, non-resectable, or metastatic urothelial carcinoma at any time prior to enrollment. Previous high grade (HG) disease is accepted as long as diagnosis date is greater than or equal to (>=5) years ago and there is documentation of low grade (LG) Ta thereafter
* Known allergies, hypersensitivity, or intolerance to any study component or its excipients
* Has a current diagnosis of newly diagnosed IR-NMIBC
* Received an investigational treatment for bladder cancer after Transurethral Resection of the Bladder Tumor (TURBT) for the current NMIBC diagnosis or within 4 weeks or the agent/therapy washout period, whichever is longer, before the planned first dose of study treatment, or is currently enrolled in an investigational study
* Evidence of current bladder perforation by cystoscopy or imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2029-07-24 (Estimated)

PRIMARY OUTCOMES:
Parts 1 to 3: Number of Participants with Adverse Events (AEs) | Up to approximately 7 years 4 months
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Parts 1 to 3: Number of Participants with AEs by Severity | Up to approximately 7 years 4 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Part 1: Number of Participants with Dose-limiting Toxicity (DLT) | Up to 28 days
  Number of participants with DLT will be assessed. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.
Part 4: Overall Complete Response (CR) in Participants with Intermediate Risk-Non-Muscle Invasive Bladder Cancer (IR-NMIBC) | Up to approximately 7 years 4 months
  Overall CR is defined as the negative cystoscopy or positive cystoscopy with centrally reviewed biopsy negative for malignancy.

SECONDARY OUTCOMES:
Parts 1 to 3: Plasma Concentration of Erdafitinib | Cohorts 1, 3 and 5: up to 6 months; Cohort 2 and 4: up to 8 weeks
  Plasma concentration of Erdafitinib will be reported.
Parts 1 to 3: Urine Concentration of Erdafitinib | Cohorts 1, 3 and 5: up to 6 months; Cohort 2 and 4: up to 8 weeks
  Urine concentration of Erdafitinib will be reported.
Parts 1 to 3: Cohorts 1 and 2: Recurrence-Free Survival (RFS) | Up to approximately 7 years 4 months
  RFS is defined as the time from start of treatment to the first detection of any new high-grade bladder cancer or upper tract urothelial carcinoma or positive urine cytology.
Parts 1 to 3: Cohort 3 and 5: Complete Response (CR) Rate | At 3 months
  CR is defined as the absence of urothelial carcinoma by cystoscopy, confirmed pathologically at first assessment, and negative urine cytology.
Parts 1 to 3: Cohort 3 and 5: Duration of CR | Up to approximately 7 years 4 months
  Duration of CR is defined as the time from first documentation of CR until the date of documented recurrence or progression, or death, whichever comes first.
Parts 1 to 3: Cohort 4: Pathological Complete Response (pCR) Rate | Up to 8 weeks
  pCR rate is defined as percentage of participants with no pathologic evidence of intravesical disease (pT0) and no pathologic evidence of nodal involvement (pN0).
Parts 1 to 3: Cohort 4: No Pathologic Evidence of Intravesical Disease (pT0) | Up to 8 weeks
  pT0 rate is defined as percentage of participants with no Pathologic Evidence of Intravesical Disease.
Parts 1 to 3: Cohort 4: Rate of downstaging to Less than (<) pT2 | Up to 8 weeks
  Rate of downstaging to <pT2 is defined as percentage of participants with pT stage <2.
Part 4: Duration of CR (DoCR) in Participants with IR-NMIBC | Up to approximately 7 years 4 months
  Duration of CR is defined as the time from first documentation of CR until the date of documented recurrence or progression, or death, whichever comes first.
Part 4: Complete Response (CR) at 3 Months in Participants with IR-NMIBC | At Month 3
  CR is defined as the negative cystoscopy or positive cystoscopy with centrally reviewed biopsy negative for malignancy at the first disease evaluation.
Part 4: Transurethral Resection of the Bladder Tumor (TURBT)-Free Survival in Participants With IR-NMIBC | Up to approximately 7 years 4 months
  Participants with TURBT-free survival will be reported.
Part 4: Number of Participants with Treatment-Emergent Adverse Event (TEAEs) by Severity | Up to approximately 7 years 4 months
  TEAEs are AEs with onset during the intervention phase or that are a consequence of a pre-existing condition that has worsened since baseline. Severity was assessed using National cancer Institute common terminology criteria for adverse events (NCI-CTCAE) version 5.0. Severity grades ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Part 4: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) Score | At baseline (Week 0), Weeks 12, 24, 36, 48, and at completion or discontinuation of study treatment (up to approximately 7 years 4 months)
  The EORTC QLQ-C30, is a self-administered, 30-item questionnaire measuring the health-related quality of life (HRQoL) of participants with cancer. EORTC QLQ-C30 includes 5 functional scales, 3 symptom scales, a global health status / quality of life scale, and 6 single items. Responses to items 1-28 are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much." Two global health status items are rated on a 7-point numeric rating scale from 1 "Very Poor" to 7 "Excellent." Higher scores indicate greater functioning, better global health status, and more severe symptoms.
Part 4: Change from Baseline in European Organization for the Research and Treatment of Cancer Non-Muscle Invasive Bladder Cancer (EORTC-QLQ-NMIBC 24) Score | At baseline (Week 0), Weeks 12, 24, 36, 48, and at completion or discontinuation of study treatment (up to approximately 7 years 4 months)
  EORTC QLQ-NMIBC24 is a 24-item questionnaire for evaluating the HRQoL of participants with non-muscle-invasive bladder cancer. The questionnaire is designed to supplement the QLQ C30 and incorporates 6 multi-item scales and 5 single items. Ratings for each item range from 1 (not at all) to 4 (very much). Higher scores indicated greater severity.
Part 4: Percentage of Participants With Clinically Meaningful Change From Baseline in EORTC-QLQ-C30 Scores | At baseline (Week 0), Weeks 12, 24, 36, 48, and at completion or discontinuation of study treatment (up to approximately 7 years 4 months)
  The EORTC QLQ-C30, is a self-administered, 30-item questionnaire measuring the HRQoL of participants with cancer. EORTC QLQ-C30 includes 5 functional scales, 3 symptom scales, a global health status/quality of life scale, and 6 single items. Responses to items 1-28 are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much." Two global health status items are rated on a 7-point numeric rating scale from 1 "Very Poor" to 7 "Excellent." Higher scores indicate greater functioning, better global health status, and more severe symptoms.
Part 4: Percentage of Participants With Clinically Meaningful Change From Baseline in EORTC-QLQ-NMIBC24 Scores | At baseline (Week 0), Weeks 12, 24, 36, 48, and at completion or discontinuation of study treatment (up to approximately 7 years 4 months)
  EORTC QLQ-NMIBC24 is a 24-item questionnaire for evaluating the HRQoL of participants with non-muscle-invasive bladder cancer. The questionnaire is designed to supplement the QLQ C30 and incorporates 6 multi-item scales and 5 single items. Ratings for each item range from 1 (not at all) to 4 (very much). Higher scores indicated greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (59):
- United States (25):
  - University of Alabama at Birmingham - The Kirklin Clinic, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - Urology Associates of Denver, Lone Tree, Colorado
  - Urological Research Network, Hialeah, Florida
  - Advanced Urology Institute, Largo, Florida
  - Advent Health Orlando, Orlando, Florida
  - Advanced Urology Institute, Oxford, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Associated Urological Specialists, Chicago Ridge, Illinois
  - Urology of Indiana, Greenwood, Indiana
  - Urologic Specialists of Northwest Indiana, Merrillville, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Southern Urology LLC, Lafayette, Louisiana
  - Greater Boston Urology, Plymouth, Massachusetts
  - Specialty Clinical Research of St Louis, St Louis, Missouri
  - Hackensack University Medical Center Urology, Hackensack, New Jersey
  - Associated Medical Professionals, Syracuse, New York
  - Levine Cancer Institute, Carolinas HealthCare System, Charlotte, North Carolina
  - Central Ohio Urology Group, Gahanna, Ohio
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Low Country Urology Clinics, North Charleston, South Carolina
  - Urology Associates, Nashville, Tennessee
  - Urology Austin, Austin, Texas
  - Urology San Antonio Research, San Antonio, Texas
- Canada (4):
  - Vancouver Prostate Centre Diamond Health Care Centre, Vancouver, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - St Josephs Healthcare Hamilton, Hamilton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Germany (7):
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - Urologicum Duisburg, Duisburg
  - Universitatsklinikum Frankfurt, Frankfurt am Main
  - Marien hospital Herne, Herne
  - Urologie Neandertal Praxis Mettmann, Mettmann
  - Universitatsklinikum Munster, Münster
  - Universitaetsklinikum Ulm, Ulm
- Israel (4):
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (4):
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Yamanashi Prefectural Central Hospital, Kofu
  - Osaka General Medical Center, Osaka
  - Toyama University Hospital, Toyama
- Netherlands (2):
  - Radboud Umcn, Nijmegen
  - UMC Utrecht, Utrecht
- South Korea (5):
  - National Cancer Center, Goyang-si
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (8):
  - Fund. Puigvert, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Reina Sofia, Córdoba
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Instituto Valenciano de Oncologia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency